CLINICAL TRIAL: NCT02681757
Title: A Comparison of Mepitel Ag vs Antibiotic Ointment When Used With the Soft Cast Technique for the Treatment of Pediatric Hand and Foot Burns, a Prospective Study
Brief Title: Comparison of Mepitel Ag vs Antibiotic Ointment Used With Soft Cast Technique for Treatment of Pediatric Burns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-1828
Record Dates: First submitted 2016-02-10; First posted 2016-02-12 (Estimated); Results first posted 2019-12-18 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Burns
Keywords: pediatric hand burn; pediatric foot burn; mepitel Ag; soft cast technique for burn wound heaing
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control- triple antibiotic ointment (Active Comparator): triple antibiotic ointment (TAO) impregnated Adaptic gauze, kling or kerlex, cast padding, gypsoma plaster, soft cast material, and coban
  Interventions: Device: triple antibiotic ointment dressing
- Variable- mepitel Ag (Experimental): mepitel Ag, kling or kerlex, cast padding, gypsoma plaster, soft cast material, and coban
  Interventions: Device: Mepitel Ag

INTERVENTIONS:
Device: triple antibiotic ointment dressing — used for control group under soft cast
  Arms: Control- triple antibiotic ointment
Device: Mepitel Ag — used for variable/experimental group under soft cast
  Arms: Variable- mepitel Ag

SUMMARY:
The aim of this study is to compare Mepitel Ag to Triple antibiotic ointment impregnated Adaptic gauze when used with the soft cast technique to assess overall time to healing, yeast infection rate and parents perception of pain level at time of dressing change on a scale of 1-10. The hypothesis is that Mepitel Ag in combination with the soft cast technique improves wound healing in pediatric partial to deep partial thickness hand and foot burns by decreasing the length of healing time, decreasing the risk of yeast infection, and decreasing pain associated with dressing changes.

DETAILED DESCRIPTION:
There is currently no gold standard dressing when it comes to treating hand or foot burns, specifically in the pediatric population. Our institution currently utilizes the soft cast technique (SCT) on all of our hand and foot burns. The SCT uses triple antibiotic ointment (TAO) impregnated Adaptic gauze, kling or kerlex, cast padding, gypsoma plaster, soft cast material, and coban. This dressing is applied one to two times during the first 2 weeks post injury. The underlying dressing is changed to nystatin impregnated Adaptic gauze, kling or kerlex, cast padding, gypsoma plaster, soft cast material, and coban for the remainder of treatment time or until surgery is indicated for debridement and grafting of wounds. The soft cast technique provides optimal positioning of the wounded hand or foot, allows for a moist wound environment, and offers protection of the injured extremity as the wound heals. The literature reveals that early surgical intervention performed in the first 7 to 10 days post injury has been shown to help achieve maximal function while decreasing the risk of hypertrophic scar formation.

A review of the current literature demonstrates silver sulfadiazine (SSD) to be the most frequently used dressing for burn wound treatment in many clinics nationwide. The use of SSD is associated with once to twice daily painful dressing changes and wound exposure that "may lead to disruption of newly formed epithelium, wound colonization, subsequent wound infection and deepening of the burn". One major benefit of the SCT is the reduction in required dressing changes, as the soft cast can stay in place for 7-10 days while maintaining optimal hand or foot positioning. This eliminates the need for painful dressing changes. Occasionally in our clinic, we have observed yeast infections under the soft cast when patients require serial casting. Other complications include occasional drying out of the adaptic gauze, which leads to painful dressing removal and interruption of the newly epithelialized wound bed. Mepitel Ag, a new soft silicone dressing produced by Molnlycke Health Care, combines Safetac technology with a silver compound to provide a broad spectrum of antimicrobial coverage, lasting up to 8 days, while minimizing damage to the new epithelium and creating a moist wound environment. The safetac technology "protects the wound and the skin. It prevents an outer dressing from sticking to the wound, therefore minimizes trauma and pain". The highly pliable nature and antimicrobial properties of the dressing make it an ideal alternative to TAO and SSD for the treatment of pediatric partial to deep partial thickness hand and foot burns.

ELIGIBILITY:
Inclusion Criteria:

* Children's Hospital Colorado burn patients
* Age 31 days to 18 years
* Newly diagnosed partial to deep partial or full thickness hand or foot burns, including bilateral or unilateral injury

Exclusion Criteria:

* silver allergy
* silicone allergy
* electrical burn
* chemical burn
* past medical history of immunodeficiency disorders such as diabetes mellitus
* h/o AIDs or HIV,
* h/o pregnant women
* prisoners
* decisionally challenged

Ages: 31 Days to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 96 (Actual)
Dates: Start 2016-09; Primary Completion 2017-09-29 (Actual); Study Completion 2017-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Moulton, M.D., Principal Investigator — University of Colorad, Childrens Hospital Colorado
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abu-Sittah GS, El Khatib AM, Dibo SA. Thermal injury to the hand: review of the literature. Ann Burns Fire Disasters. 2011 Dec 31;24(4):175-85. PMID 22639560
- [Background] Barret JP, Herndon DN. Plantar burns in children: epidemiology and sequelae. Ann Plast Surg. 2004 Nov;53(5):462-4. doi: 10.1097/01.sap.0000136973.62109.cf. PMID 15502462
- [Background] Briggs SL, Taylor A, Lansdown AB. Clinical perspective on silicone dressings and wound management. J Wound Care. 2008 Aug;17(8):364-5; author reply 365-6. doi: 10.12968/jowc.2008.17.8.30801. No abstract available. PMID 18754199
- [Background] Brown M, Dalziel SR, Herd E, Johnson K, Wong She R, Shepherd M. A Randomized Controlled Study of Silver-Based Burns Dressing in a Pediatric Emergency Department. J Burn Care Res. 2016 Jul-Aug;37(4):e340-7. doi: 10.1097/BCR.0000000000000273. PMID 26171678
- [Background] Bugmann P, Taylor S, Gyger D, Lironi A, Genin B, Vunda A, La Scala G, Birraux J, Le Coultre C. A silicone-coated nylon dressing reduces healing time in burned paediatric patients in comparison with standard sulfadiazine treatment: a prospective randomized trial. Burns. 1998 Nov;24(7):609-12. doi: 10.1016/s0305-4179(98)00095-3. PMID 9882058
- [Background] Choi M, Armstrong MB, Panthaki ZJ. Pediatric hand burns: thermal, electrical, chemical. J Craniofac Surg. 2009 Jul;20(4):1045-8. doi: 10.1097/scs.0b013e3181abb25f. PMID 19634213
- [Background] Duteille F, Jeffery SL. A phase II prospective, non-comparative assessment of a new silver sodium carboxymethylcellulose (AQUACEL((R)) Ag BURN) glove in the management of partial thickness hand burns. Burns. 2012 Nov;38(7):1041-50. doi: 10.1016/j.burns.2012.05.001. Epub 2012 Jun 5. PMID 22677163
- [Background] Feldmann ME, Evans J, O SJ. Early management of the burned pediatric hand. J Craniofac Surg. 2008 Jul;19(4):942-50. doi: 10.1097/SCS.0b013e318175f38d. PMID 18650716
- [Background] Gee Kee E, Kimble RM, Cuttle L, Stockton K. Comparison of three different dressings for partial thickness burns in children: study protocol for a randomised controlled trial. Trials. 2013 Nov 25;14:403. doi: 10.1186/1745-6215-14-403. PMID 24274190
- [Background] Johnson J, Silverberg R. Serial casting of the lower extremity to correct contractures during the acute phase of burn care. Phys Ther. 1995 Apr;75(4):262-6. doi: 10.1093/ptj/75.4.262. PMID 7899484
- [Background] Meuleneire F, Rucknagel H. Soft Silicone dressings made easy. Wounds International 2013.
- [Background] Mitura K, Oslowska J, Mitura A. A Change of Traditional Method of Treatment of Partial Thickness Burn with Hydrofibre Dressings. Pol Przegl Chir. 2015 Feb;87(2):91-6. doi: 10.1515/pjs-2015-0025. PMID 26146101
- [Background] White R, Morris C. Mepitel: a non-adherent wound dressing with Safetac technology. Br J Nurs. 2009 Jan 8-21;18(1):58-64. doi: 10.12968/bjon.2009.18.1.93582. PMID 19127235
- [Background] Toussaint J, Chung WT, Osman N, McClain SA, Raut V, Singer AJ. Topical antibiotic ointment versus silver-containing foam dressing for second-degree burns in swine. Acad Emerg Med. 2015 Aug;22(8):927-33. doi: 10.1111/acem.12723. Epub 2015 Jul 22. PMID 26202791

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control- Triple Antibiotic Ointment | Variable- Mepitel Ag
Started | 47 | 49
Completed | 47 | 49
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control- Triple Antibiotic Ointment | Variable- Mepitel Ag | Total
Number analyzed (Participants) | 47 | 49 | 96
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 47 | 49 | 96
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 2.3 [1.3 to 6.5] | 1.6 [1.1 to 3.0] | 1.8 [1.1 to 6.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 15 | 35
  Male | 27 | 34 | 61
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 47 | 49 | 96

OUTCOME MEASURES:

1. Primary Outcome: Change in Wound Appearance From Initial Injury Until Wound Healed
Description: Burn will be evaluated every 3-7 days from date of randomization for up to 21 days (End of Study) after application of Mepitel Ag or triple antibiotic ointment impregnated Adaptic gauze to determine if the burn healed or not.
Time Frame: Up to 21 days
Population: Some participants had multiple burns. We investigated all burns.
Measure: Count of Units; unit: Burns
Units Other Than Participants: Burns
Arm/Group | Control- Triple Antibiotic Ointment | Variable- Mepitel Ag
Number analyzed (Participants) | 47 | 49
Number analyzed (Burns) | 53 | 60
Burns | 43 | 51

2. Secondary Outcome: Evaluation of Pain Level
Description: Subject will be evaluated at first post-operative follow up visit ranging from date of surgery up to 21 days (End of Study) for level of pain at time of dressing change based on FLACC scale and calculated per Nurse and parent perceived level of patient pain. "The Face, Legs, Activity, Cry, Consolability scale or FLACC scale is a measurement used to assess pain for children between the ages of 2 months and 7 years or individuals that are unable to communicate their pain. The scale is scored in a range of 0-10 with 0 representing no pain. The scale has five criteria, which are each assigned a score of 0, 1 or 2."
Time Frame: Up to 21 days from date of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Control- Triple Antibiotic Ointment | Variable- Mepitel Ag
Number analyzed (Participants) | 47 | 49
Participants
  0 | 31 | 24
  1 | 6 | 7
  2 | 0 | 7
  3 | 2 | 1
  4 | 1 | 2
  5 | 2 | 0
  6 | 1 | 2
  7 | 2 | 0
  8 | 0 | 1
  Not Reported | 2 | 5

3. Secondary Outcome: Presence of Yeast Infection in Burn Wound
Description: Subject will be evaluated every 3-7 days from date of randomization for up to 21 days (End of Study) for clinically observed evidence of yeast infection from visible wound inspection at time of dressing change, i.e.: foul yeast odor, red erythematous rash.
Time Frame: Up to 21 days
Population: The unit of observation is a single burn, not an individual patient. This outcome is number of yeast infections per burn dressing group.
Measure: Number; unit: burns
Units Other Than Participants: Burns
Arm/Group | Control- Triple Antibiotic Ointment | Variable- Mepitel Ag
Number analyzed (Participants) | 47 | 49
Number analyzed (Burns) | 53 | 60
burns | 5 | 6

ADVERSE EVENTS:
Time Frame: 15 months
Arm/Group | Control- Triple Antibiotic Ointment | Variable- Mepitel Ag
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/49
Other Adverse Events (participants affected / at risk) | 0/47 | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-08): https://cdn.clinicaltrials.gov/large-docs/57/NCT02681757/Prot_SAP_000.pdf